CLINICAL TRIAL: NCT00071266
Title: The Dose Response of Niacin ER/Lovastatin on Peak Walking Time (PWT) in Patients With Intermittent Claudication - a Matrix Design
Brief Title: The Dose Response of Niacin ER/Lovastatin on Peak Walking Time (PWT) in Patients With Intermittent Claudication - TROPIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kos Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MA-03-010401; The TROPIC Study
Record Dates: First submitted 2003-10-16; First posted 2003-10-20 (Estimated); Last update posted 2006-11-02 (Estimated); Status verified 2006-10

CONDITIONS: Intermittent Claudication; Peripheral Vascular Disease
Keywords: Intermittent Claudication; Peripheral Arterial Disease; Atherosclerosis; Niacin; Lovastatin; PAD; IC
MeSH Terms: conditions — Intermittent Claudication; Peripheral Vascular Diseases; Peripheral Arterial Disease; Atherosclerosis | interventions — Lovastatin

INTERVENTIONS:
Drug: Niacin Extended Release and Lovastatin Tablets

SUMMARY:
The purpose of this study is to compare the dose response and safety of Niacin ER/Lovastatin, Niaspan® and Lovastatin with each other, in subjects with leg pain caused by a narrowing of their leg arteries.

At least 870 subjects, with leg pain caused by a narrowing of their leg arteries will take part in this study.

Both Niaspan and lovastatin (Mevacor®) are approved by the United States Food and Drug Administration (FDA) to treat high cholesterol. Niacin ER/Lovastatin (Advicor®), a combination of these two drugs, is also approved by the FDA to treat high cholesterol. The use of Niacin ER/Lovastatin to treat narrowing of leg arteries and relieve "intermittent claudication" (leg pain caused by narrowing of the arteries in the leg) is considered investigational. An investigational use is one that is not approved by the FDA.

DETAILED DESCRIPTION:
This is a Phase 3, 32-week, double-blind, diet-intervention, randomized, parallel group, ten-arm, multi-center, multi-national, dose titration study evaluating the safety and efficacy of NL in patients with intermittent claudication (IC).

The objectives of this study are to evaluate the safety and efficacy of NL in patients with IC. The primary efficacy analysis will be the percent change from baseline in Peak Walking Time (PWT) calculated from the natural logarithm of the ratio of the time walked on treadmill at the Week 32 Visit divided by the time walked at baseline. Other efficacy measures will include Claudication Onset Time (COT) percent changes from baseline to Week 32 , changes in Ankle Brachial Index (ABI), Quality of Life (QoL) percent changes at Weeks 20 and 32, lower limb amputations, composite of cardiovascular events (MI, stroke, and vascular death), and coronary and peripheral artery revascularizations. Safety variables will include serum transaminases, routine chemistry parameters, hematology, and adverse events. Pharmacokinetic analyses will be conducted as well.

ELIGIBILITY:
INCLUSION CRITERIA:

* Men & women at least 40 years of age or older. Women must not be pregnant nor breast-feeding & not planning to become pregnant or to breast-feed.
* History of IC of the lower extremities which has been present for at least 6 months with no change in symptoms in the previous 3 months prior to screening.
* LDL-C of <160 mg/dL and Triglycerides <800.

EXCLUSION CRITERIA:

* Severe neuropathy.
* Gross obesity (BMI ≥ 40).
* Presence of critical limb ischemia defined as ischemic rest pain, gangrene, ulceration, or pending amputation of a lower extremity due to severe PAD.
* Surgical intervention to alleviate symptoms of claudication within 6 months or endovascular interventions within 3 months.
* Documented CAD taking any cholesterol-modifying agent and unable to undergo washout as judged by the Investigator or due to personal choice.
* Systolic blood pressure ≥160 mmHg &/or diastolic blood pressure ≥95 mmHg.
* Presence of clinically significant laboratory test abnormalities for liver or renal function tests, thyroid function or HgbA1C.
* History of alcohol abuse or currently drinks alcohol in excess.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 870
Dates: Start 2003-10

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Tatum Ridge Internal Medicine, Phoenix, Arizona
  - Scottsdale Cardiovascular Research Institute, LLC, Scottsdale, Arizona
  - VA Palo Alto Health Care System, Palo Alto, California
  - University of California-Davis; Department of Surgery, Sacramento, California
  - Sacramento Heart & Vascular Medical Associates, Sacramento, California
  - Clinical Research Center of California, San Diego, California
  - North County Internal Medicine, Vista, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Cardiovascular Center of Sarasota, Sarasota, Florida
  - Clinical Research Center of Georgia, Warner Robins, Georgia
  - River Cities Cardiology, MPC, Jeffersonville, Indiana
  - HPV Heart P.A., Columbia, Maryland
  - St. Joseph Mercy-Oakland Research Office, Pontiac, Michigan
  - Saint Louis University, St Louis, Missouri
  - Carolina Pharmaceutical Research, Statesville, North Carolina
  - COR Clinical Research, Oklahoma City, Oklahoma
  - New Hope Research of Oregon, Portland, Oregon
  - Penn State College of Medicine, Hershey, Pennsylvania
  - Radiant Research, Philadelphia, Pennsylvania
  - Mainline Health Heart Center, Wynnewood, Pennsylvania
  - Clinical Cardiology Research Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Pro Research Group, LLC, San Antonio, Texas
  - Hampton Roads Center for Clinical Research, Inc., Norfolk, Virginia
  - Care Foundation, Inc, Wausau, Wisconsin